CLINICAL TRIAL: NCT05859217
Title: A Multi-center Phase II Study of Combining Cabozantinib and Atezolizumab as the 1st Line Therapy for PD-L1 Negative Advanced/Metastatic NSCLC (Cabatezo-1)
Brief Title: A Study of Combining Cabozantinib and Atezolizumab for Advanced/Metastatic NSCLC (Cabatezo-1)
Acronym: Cabatezo-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jun Zhang, MD, PhD (Other)
Collaborators: Exelixis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, MD, PhD, Associate Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2021-Cabatezo-1
Record Dates: First submitted 2023-02-18; First posted 2023-05-15 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer; NSCLC Stage IV; Metastatic NSCLC - Non-Small Cell Lung Cancer; Advanced NSCLC
Keywords: Cancer immunotherapy; anti-angiogenesis; Investigator-initiated clinical trial
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib and Atezolizumab (Experimental): Cabozantinib 40mg po daily + Atezolizumab 1200mg iv on day 1; 1 cycle = 21 days
  Interventions: Drug: Cabozantinib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Cabozantinib — Oral once per day, Days 1 - 21 every 21 days
  Other Names: Cabometyx
Drug: Atezolizumab — Intravenous (IV) once every 21 days
  Other Names: Tecentriq

SUMMARY:
NSCLC patients with low expression level of PD-L1, esp. those with its level less than 1%, do not derive much benefit from anti-PD-1/L1 therapy (e.g. atezoilzumab). In this study, investigators hypothesize that the combination of cabozantinib (a multi-kinase inhibitor) and atezolizumab will result in better therapeutic value.

DETAILED DESCRIPTION:
For metastatic/advanced non-small cell (NSCLC) patients who do not have targetable mutations, the combination of chemotherapy with immunotherapy targeting the programmed death-1 and its ligand (PD-1/L1) is now a standard of care. In addition, recent studies also demonstrated that immunotherapy doublet using anti-PD-1 agent nivolumab and anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) agent ipilimumab could be another valid option. However, largely due to the immunosuppressive tumor microenvironment, the therapeutic response remains suboptimal in NSCLC patients with PD-L1 tumor proportion score (TPS) lower than 1% (aka PD-L1 negative). For example, the objective response rate (ORR) in KEYNOTE-189 was 32.3% using pembrolizumab plus chemotherapy, and only 27.3% in Checkmate 227 study using nivolumab and ipilimumab, in the PD-L1 negative population. These observations necessitate the search for novel combinations to benefit our PD-L1 negative NSCLC patients.

The investigators hypothesize that the combination of cabozantinib and atezolizumab is such an innovative strategy based on the following rationales: 1) cabozantinib is a multi-kinase inhibitor, and some of the targets, for example the vascular endothelial growth factor (VEGF) pathway is notorious to confer immune suppressive tumor microenvironment. In fact, our previous study has demonstrated that anti-VEGF synergizes anti-PD-1 in preclinical model. Consistent with this, cabozantinib has been shown to increase tumor infiltrative cytotoxic CD8+ T cells, reduce immune suppressive T regulatory cells (Tregs) and myeloid-derived suppressor cells (MDSCs), as well as activate anti-tumor innate immunity in multiple solid tumors; 2) at the animal level, cabozantinib was found synergistic with anti-PD-1 agents to elicit anti-tumor immune response; and 3) more importantly, at the human level, the combination of cabozantinib with atezolizumab was found safe in Cohort 7 of the phase 1b COSMIC-021 study and achieved 27% ORR in previously immunotherapy-treated NSCLC - suggesting a potentially higher efficacy if such combination is to be used in the 1st line setting.

The investigators therefore propose here the combination of cabozantinib and atezolizumab to be used as the 1st line treatment for advanced/metastatic NSCLC with negative PD-L1 expression.

ELIGIBILITY:
INCLUSION CRITERIA:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Males and females age ≥ 18 years
* ECOG Performance Status 0 - 1
* Pathologically confirmed advanced/metastatic NSCLC, with PD-L1<1% based on IHC using 22C3 antibody
* At least one target lesion that can be assessed by RECIST 1.1
* For candidates who are not qualified for upfront FDA-approved targeted therapy, must be systemic treatment naïve (local palliative RT more than 4 weeks prior is allowed)
* For candidates who are qualified for upfront FDA-approved targeted therapy (e.g. having sensitizing mutations in EGFR, ALK and BRAF, etc.), treatment must have failed and received at least one line of ONLY FDA-approved targeted therapy
* Availability of a representative tumor specimen for correlative research. Optional but highly recommended: willing to undergo tumor tissue biopsy only if deemed safe and feasible by the investigator.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
* Women of childbearing potential must have a negative serum pregnancy test 72 hours prior to initiating treatment. Female participants are considered to be of childbearing potential unless one of the following criteria is met: documented permanent sterilization (hysterectomy, bilateral salpingectomy, or bilateral oophorectomy) or documented postmenopausal status (defined as 12 months of amenorrhea in a woman > 45 years-of-age in the absence of other biological or physiological causes. In addition, females < 55 years-of-age must have a serum follicle stimulating (FSH) level > 40 mIU/mL to confirm menopause). Note: Documentation may include review of medical records, medical examinations, or medical history interview by study site.
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use two forms of adequate contraception (hormonal AND barrier method of birth control) prior to study entry, for the duration of study participation and for 6 months following completion of therapy.
* Men of child-bearing potential must not father a child or donate sperm while on this study and for 6 months after the last study treatment.
* Adequate organ function
* Negative HIV test at screening, with the following exception: patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count >200/uL, and have an undetectable viral load. They must agree to continue on such anti-retroviral therapy per local standard treatment guideline
* Negative HBV and HCV tests at screening, with the following exception:

  * For HBV: DNA must be < 500 IU/mL (or must be < 2500 copy/mL if copy/mL is the only unit available in the study site; if the normal ranges of the study sites are different, the positive standard must not be met), and have received anti-HBV therapy for at least 14 days prior to the first dose of study treatment (treatment in accordance with local standard of care, e.g., entecavir) and are willing to receive antiviral therapy throughout the study if indicated;
  * For HCV (with positive HCV RNA): must receive anti-viral therapy in accordance with the local standard treatment guideline and hepatic function resolve to CTCAE Grade ≤1

EXCLUSION CRITERIA:

* Simultaneously enrolled in any therapeutic clinical trial
* Current or anticipating use of other investigational agents while participating in this study
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Diagnosed with a psychiatric illness or is in a social situation that would limit compliance with study requirements
* Active Grade 3 (per the NCI CTCAE, Version 5.0) or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment
* Patients harboring targetable mutations (e.g., EGFR, ALK and BRAF, etc.) who have not had at least one frontline targeted therapy fail, or have received other systemic therapies (e.g. chemotherapy, immunotherapy, etc.)
* Patients with carcinomatous meningitis (leptomeningeal metastasis)
* Undergone major surgery within 2 weeks prior to the start of study regimen, or has not achieved complete wound healing
* Presence of another cancer with disease manifestations or therapy that could adversely affect participant safety or longevity, create the potential for drug-drug interactions, or compromise the interpretation of study results. Otherwise, patients can be considered eligible, for example, locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Prior treatment with cabozantinib and/or atezolizumab.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment
* Radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before first dose of study treatment. Participants with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks prior to first dose of study treatment after radiotherapy or at least 4 weeks prior to first dose of study treatment after major surgery (e.g., removal or biopsy of brain metastasis). Participants must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Eligible participants must be neurologically asymptomatic and with corticosteroid no more than 10mg prednisone or equivalent at the time of first dose of study treatment.
* Concomitant anticoagulation with coumarin agents (e.g., warfarin), direct thrombin inhibitors (e.g., dabigatran), direct factor Xa inhibitor betrixaban, or platelet inhibitors (e.g., clopidogrel). Allowed anticoagulants are the following:

  * Prophylactic use of low-dose aspirin for cardio-protection (per local applicable guidelines) and low-dose low molecular weight heparins (LMWH).
  * Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors such as rivaroxaban, edoxaban, or apixaban in participants without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before first dose of study treatment without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.
* Live, attenuated vaccines (e.g., FluMist) are prohibited within 4 weeks prior to initiation of study treatment, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab.
* The participant has uncontrolled, significant cardiovascular disorders
* Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (e.g., pulmonary hemorrhage) within 12 weeks before first dose of study treatment
* Lesions invading or encasing any major blood vessels.
* Other clinically significant disorders that would preclude safe study participation
* Major surgery (e.g., laparoscopic nephrectomy, GI surgery, removal or biopsy of brain metastasis) within 2 weeks before first dose of study treatment. Minor surgeries within 10 days before first dose of study treatment. Participants must have complete wound healing from major surgery or minor surgery before first dose of study treatment. Participants with clinically relevant ongoing complications from prior surgery are not eligible
* Pregnant or lactating females.
* Inability to swallow tablets or unwillingness or inability to receive IV administration.
* Previously identified allergy or hypersensitivity to Chinese hamster ovary cell products, or components of the study treatment formulations or history of severe infusion-related reactions to monoclonal antibodies.
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
* Active or history of autoimmune disease or immune deficiency (see Appendix I), including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Any serious illness, uncontrolled inter-current illness, psychiatric illness, active or uncontrolled infection, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with the patient's participation in the study, or with the interpretation of the results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 1 year
  From baseline to End of Treatment (EOT) due to disease progression using RECIST criteria 1.1

SECONDARY OUTCOMES:
Duration of response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The response to the study drugs will be determined using RECIST criteria 1.1
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  The lack of progression will be dertermined using RECIST criteria 1.1
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Medical Record will be followed to watch survival status
Drug Safety | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Safety of drugs will be determined by documenting adverse events and the severity of adverse events will be documented using CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Study Chair — University of Kansas Medical Center
Locations (4):
- United States (4):
  - The University of Kansas Cancer Center - Westwood, Kansas City, Kansas
  - The University of Kansas Cancer Center - Indian Creek, Overland Park, Kansas
  - The University of Kansas Cancer Center - North, Kansas City, Missouri
  - The University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri